CLINICAL TRIAL: NCT05391464
Title: Preoperative Versus Postoperative Peripheral Nerve Block for Pain Control After Ankle and Wrist Fracture Surgery
Brief Title: Nerve Block for Pain Control After Fracture Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MaineGeneral Health (Other)
Responsible Party: Principal Investigator, Stuart A Aitken, Principal Investigator, MaineGeneral Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNBtrial
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Ankle Fractures; Distal Radius Fracture
MeSH Terms: conditions — Ankle Fractures; Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Randomized, single-center, superiority
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripheral Nerve Block (Active Comparator): Participants will receive an ultrasound-guided, single shot PNB using 30ml 0.5% bupivacaine with 10mg dexamethasone. The anatomic location of the block will be determined by the anesthesiologist and will vary according to fracture location and anticipated surgical approaches. Intraoperative sedation will be used at the discretion of the anesthetic team.
  Interventions: Procedure: Peripheral Nerve Block
- General Anesthesia +/- PNB (Active Comparator): GA will be administered in the operating room by a nurse anesthetist, with support from the anesthesiologist. GA will be induced with propofol and fentanyl and maintained with sevoflurane or desflurane and fentanyl. Doses will be determined by the anesthesiology team.
  Interventions: Procedure: Peripheral Nerve Block

INTERVENTIONS:
Procedure: Peripheral Nerve Block — Utilized preoperatively with sedation during surgery, or postoperatively for additional anesthesia after GA.

SUMMARY:
Surgical treatment for patients with a fracture of the ankle or distal radius is commonly offered on an outpatient basis. Patients are routinely discharged from hospital within 4 hours of their procedure. The surgery is commonly performed under peripheral nerve block with sedation, or under general anesthesia with postoperative peripheral nerve block, (if required for analgesic purposes). It is unclear which of these two strategies offers patients superior pain relief in the first few days following surgery. This trial aims to compare the pain intensity and analgesic medication consumption between patients in these two groups.

DETAILED DESCRIPTION:
Background:

Open reduction and internal fixation (ORIF) surgery for a fracture of the ankle or distal radius is a commonly performed outpatient orthopedic procedure. Surgery is routinely performed under a preoperative peripheral nerve block (PNB) with sedation, or under general anesthesia (GA) with supplemental postoperative PNB for analgesic purposes. The method chosen is often influenced by the opinion and experience of the anesthetic team. There is no consensus as to whether PNB should be utilized preoperatively, or reserved for 'as needed' cases postoperatively.

The use of PNB in fracture surgery has been recommended in order to reduce perioperative opioid analgesic requirements and improve postoperative pain, particularly in the context of the ongoing opioid epidemic. For patients undergoing ORIF for ankle or distal radius fractures, successfully administered PNB can provide excellent pain relief in the first 8 to 12 hours post-surgery. However, a concern with PNB is rebound pain, the presence of delayed acute postoperative pain at 12 to 24 hours, affecting up to 50% of patients.

With a majority of extremity fracture surgeries performed on an outpatient basis, patients who experience rebound pain will do so after leaving hospital. PNB might therefore not provide satisfactory analgesia when patients are in most need of it. Instead, GA might offer a more desirable postoperative pain profile with patients experiencing peak pain intensity shortly after surgery, followed by steady improvement prior to discharge. In the context of rationalizing the potency of discharge prescription opioids, having less pain post-discharge is preferable.

Rather than universally adopting preoperative PNB for those undergoing ankle or distal radius ORIF, a more targeted approach might improve patients' postoperative pain experience. Performing surgery under GA, and offering postoperative PNB 'as needed' to those whose pain is poorly controlled, has the advantage of avoiding the risks of PNB administration (and potential post-discharge rebound pain) in patients whose pain is manageable after GA. Furthermore, while preoperative PNB is associated with decreased intraoperative opioid requirement, there is no consensus that offering PNB postoperatively is clinically inferior in terms of the analgesia provided, or the subsequent risk of rebound pain.

Primary Aim:

The primary aim of the trial is to determine if any difference exists between (1) preoperative PNB and (2) GA with 'as needed' postoperative PNB with respect to the primary outcome measure, reported pain intensity (0-10, visual analogue scale), at 24 hours post-surgery for adult patients undergoing ORIF for a fracture of the ankle or distal radius.

Secondary Aims:

The secondary aims include determining if a difference exists between groups with regards to pain at discharge, pain 12 hours post-surgery, pain at 48 hours, pain at 72 hours. In addition, the functional activity scale and analgesic consumption (opioid plus nonopioid) will be compared at these time points.

Methodology:

Single-center, prospective, randomized, open label, superiority trial including adult patients receiving surgery for an acute, isolated, fracture of either the ankle or distal radius.

The minimum clinically important difference for pain, as reported in the pain literature, is 1.5 to 2 points on an eleven-point (0 to 10) visual analogue scale. An a priori power analysis determined that 68 participants would provide sufficient power to detect a difference in mean pain scores of 1.5 or more between trial groups, assuming a standard deviation of 2.2 points (alpha 0.05, 80% power).

Suitable patients will be recruited from the outpatient orthopedic clinic. Participants will be randomized to one of two groups for each fracture type (ankle and wrist) using 3 blocks of sealed study envelopes: "PNB" or "GA+/-PNB". They will then be scheduled on the next available OR list as either the first or second case to allow time for postoperative data capture. Routine postoperative prescriptions will be sent electronically to the pharmacy and participants will be given written trial material to take home and review.

Willingness to participate in the trial will be confirmed on the day of surgery, and the method of anesthesia confirmed with the anesthesiologist and nurse anesthetist. Following surgery, PNB patients will return to the Day Surgery Unit (DSU) and GA patients will be taken to the Post Anesthesia Care Unit (PACU). Standard analgesia will be administered to both groups as part of routine care.

GA patients whose pain is poorly controlled despite multiple doses of short-acting opioid will be offered PNB postoperatively. This postoperative PNB will be administered at the discretion of the PACU team and anesthesiologist.

Pain scores and analgesic consumption will be recorded for each trial participant prior to discharge from hospital. A contact telephone number will be confirmed.

The participant will be contacted by telephone to obtain outcome data at 12 hours (evening of surgery), 24 hours (following morning), at 48 hours and at 72 hours. During each call, patients will be routinely counseled about postoperative pain management. All other office follow-up visits will be competed as part of routine.

ELIGIBILITY:
Inclusion Criteria:

* Within 2 weeks of injury
* Isolated fracture requiring surgery
* Outpatient

Exclusion Criteria:

* Multiple fractures
* Inpatients
* Cognitive impairment
* Unable to comply with follow-up
* No means of telephone contact
* Contraindication to peripheral nerve block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-05-18 (Estimated); Study Completion 2025-06-18 (Estimated)

PRIMARY OUTCOMES:
Pain 24 hours | 24 hours postop
  Patient-rated measure, 0-10 visual analogue scale

SECONDARY OUTCOMES:
Pain 12 hours | 12 hours postop
  0-10 visual analogue scale
Nausea and Vomiting 24 hours | 24 hours postop
  0-10 visual analogue scale
Pain Functional Activity Scale 24 hours | 24 hours postop
  A - No limitation, minimal pain; B - Mild limitation, moderate to severe pain; C - Severe limitation, can't perform due to severe pain. Four domains: Getting dressed, Preparing food, Moving around, Sleeping
Pain Functional Activity Scale 48 hours | 48 hours postop
  A - No limitation, minimal pain; B - Mild limitation, moderate to severe pain; C - Severe limitation, can't perform due to severe pain. Four domains: Getting dressed, Preparing food, Moving around, Sleeping
Pain 48 hours | 48 hours postop
  0-10 visual analogue scale

OTHER OUTCOMES:
Analgesic consumption | 24 hours, 48 hours, 72 hours postop
  Total milligram morphine equivalents, and nonopioid analgesics
Rebound pain | First 72 hours postop
  Proportion of participants experiencing rebound pain (defined as visual analogue scale pain of 3 or less, climbing to 7 or more) after PNB.

CONTACTS AND LOCATIONS:
Locations (1):
- MaineGeneral Medical Center, Augusta, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barry GS, Bailey JG, Sardinha J, Brousseau P, Uppal V. Factors associated with rebound pain after peripheral nerve block for ambulatory surgery. Br J Anaesth. 2021 Apr;126(4):862-871. doi: 10.1016/j.bja.2020.10.035. Epub 2020 Dec 31. PMID 33390261
- [Background] Fang J, Shi Y, Du F, Xue Z, Cang J, Miao C, Zhang X. The effect of perineural dexamethasone on rebound pain after ropivacaine single-injection nerve block: a randomized controlled trial. BMC Anesthesiol. 2021 Feb 12;21(1):47. doi: 10.1186/s12871-021-01267-z. PMID 33579199
- [Background] Galos DK, Taormina DP, Crespo A, Ding DY, Sapienza A, Jain S, Tejwani NC. Does Brachial Plexus Blockade Result in Improved Pain Scores After Distal Radius Fracture Fixation? A Randomized Trial. Clin Orthop Relat Res. 2016 May;474(5):1247-54. doi: 10.1007/s11999-016-4735-1. Epub 2016 Feb 11. PMID 26869374
- [Background] Goldstein RY, Montero N, Jain SK, Egol KA, Tejwani NC. Efficacy of popliteal block in postoperative pain control after ankle fracture fixation: a prospective randomized study. J Orthop Trauma. 2012 Oct;26(10):557-61. doi: 10.1097/BOT.0b013e3182638b25. PMID 22732860
- [Background] Hsu JR, Mir H, Wally MK, Seymour RB; Orthopaedic Trauma Association Musculoskeletal Pain Task Force. Clinical Practice Guidelines for Pain Management in Acute Musculoskeletal Injury. J Orthop Trauma. 2019 May;33(5):e158-e182. doi: 10.1097/BOT.0000000000001430. PMID 30681429
- [Background] Kanto K, Lahdeoja T, Paavola M, Aronen P, Jarvinen TLN, Jokihaara J, Ardern CL, Karjalainen TV, Taimela S. Minimal important difference and patient acceptable symptom state for pain, Constant-Murley score and Simple Shoulder Test in patients with subacromial pain syndrome. BMC Med Res Methodol. 2021 Mar 6;21(1):45. doi: 10.1186/s12874-021-01241-w. PMID 33676417
- [Background] Laigaard J, Pedersen C, Ronsbo TN, Mathiesen O, Karlsen APH. Minimal clinically important differences in randomised clinical trials on pain management after total hip and knee arthroplasty: a systematic review. Br J Anaesth. 2021 May;126(5):1029-1037. doi: 10.1016/j.bja.2021.01.021. Epub 2021 Mar 5. PMID 33678402
- [Background] Richebe P, Rivat C, Liu SS. Perioperative or postoperative nerve block for preventive analgesia: should we care about the timing of our regional anesthesia? Anesth Analg. 2013 May;116(5):969-970. doi: 10.1213/ANE.0b013e31828843c9. No abstract available. PMID 23606468